CLINICAL TRIAL: NCT00215683
Title: An Open-Label, Multi-Centre, Extension Study Evaluating the Long-Term Safety and Tolerability of Degarelix One-Month Depots in Patients With Prostate Cancer.
Brief Title: An Extension Study Evaluating the Long-Term Safety and Tolerability of Degarelix One-Month Depots in Prostate Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS12A
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2010-12-14 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen ablation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Degarelix 80 mg (Experimental): Participants who completed the CS12 study in the Degarelix 80 mg arm continued that dose into the CS12A extension study. After a protocol amendment in January 2006 all study participants were treated with 160 mg (40 mg/mL).
  Interventions: Drug: Degarelix
- Degarelix 120 mg (Experimental): Participants who completed the CS12 study in the Degarelix 120 mg arm continued that dose into the CS12A extension study. After a protocol amendment in January 2006 all study participants were treated with 160 mg (40 mg/mL).
  Interventions: Drug: Degarelix
- Degarelix 160 mg (Experimental): Participants who completed the CS12 study in the Degarelix 160 mg arm continued that dose into the CS12A extension study. After a protocol amendment in January 2006 all study participants were treated with 160 mg (40 mg/mL).
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Drug supplied as a powder to be dissolved in the solvent for solution for injection. Degarelix given by subcutaneous injection every 28 days until the end of the study.
  Other Names: Degarelix acetate; FE200486

SUMMARY:
This was an extension study for the study FE200486 CS12 (NCT00819156). Each participant was to be treated until he was discontinued or withdrawn from the study, or a marketing authorization for degarelix had been obtained.

The study was terminated when all ongoing participants had been treated for at least 5 years (including one year in the main study).

DETAILED DESCRIPTION:
Participants who completed the main FE200486 CS12 study initially continued with the same dose in the FE200486 CS12A extension study. After a protocol amendment all study participants were treated with 160 mg (40 mg/mL).

The data include data from the participants who participated in both the main study (FE200486 CS12; NCT00819156) and the extension study FE200486 CS12A.

ELIGIBILITY:
Inclusion criteria:

* Had given written consent before any study-related activity was performed (a study-related activity was defined as any procedure that would not have been performed during the normal management of the participant)
* Had completed the FE200486 CS12 study

Exclusion criterion:

* Had been withdrawn from the FE200486 CS12 study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2005-02; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (34):
- Belgium (3):
  - UCL Saint Luc, Brussels
  - UZ Gent, Ghent
  - UZ Gasthuisberg, Urology Department, Leuven
- Germany (2):
  - Vivantes Klinikum am Urban, Klinik für Urologie, Berlin
  - Urologische Universitätsklinikum, Klinikum Mannheim GmbH, Fakultät für Klinische Medizin Mannheim, Mannheim
- Hungary (7):
  - Bajcsy-Zsilinszky Hospital, of local Government of Budapest, Dept. of Urology, Budapest
  - Jahn Ferenc Dél-Pesti Hospital, Dept. of Urology, Budapest
  - Pez Aladar County Hospital, Dept. of Urology, Győr
  - Bács-Kiskun County Hospital, Dept. of Urology, Kecskemét
  - BAZ County Hospital, Dept of Urology, Miskolc
  - Hospital of Local Government of Szeged, Dept. of Urology, Szeged
  - MÁV Hospital, Dept. of Urology, Szolnok
- Netherlands (2):
  - Academic Medical Center, Dept. of Urology, Amsterdam
  - Atrium MC, Dept. of Urology, Heerlen
- Romania (4):
  - "Prof.Dr.Th.Burghele" Hospital - Bucharest, Bucharest
  - "Sf. Ioan" Emergency Hospital - Urology Department, Bucharest
  - CF2 Hospital - Bucharest, Urology Department, Bucharest
  - Fundeni Clinical Institute - Bucharest, Urology Department, Bucharest
- Russia (11):
  - Moscow State University of Medicine and Dentistry, Department of Urology, Urogynecology and Andrology, City Hospital #50, Urology Department, Moscow
  - Russian Medical Academy of Postgraduate Education, Department of Gerontolology and Geriatrics, Moscow City Hospital #60, Urology Department, 84/1, Entuziastov Shosse (Hospital), Moscow
  - Russian Medical Academy of Postgraduate Education, Urology Department, Moscow Clinical Hospital n.a. Botkin, Urology Department, 5/16, 2-oy Botkinsky proezd (Hospital), Moscow
  - Russian State Medical University, Department of Urology and Surgical Nephrology, Moscow City Hospital #1, Moscow
  - "Andros" Urology Clinic, 36A, Lenina St., Saint Petersburg
  - City Hospital #15, Urology Department, Saint Petersburg
  - City Hospital #26, Urology Department, Saint Petersburg
  - I.I. Mechnikov St. Petersburg State Medical Academy, Urology Department, Saint Petersburg
  - Research Institute of Urology of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - St. Petersburg Pavlov Medical School, Urology Department, Saint Petersburg
  - St.Petersburg Pavlov Medical School, Outpatient Diagnostic Center, Saint Petersburg
- South Africa (5):
  - Glenwood Hospital, Durban
  - WITS Medical School, Level 9, Parktown
  - 401 B Medical Centre, Pietermaritzburg
  - Pretoria Urology Hospital, Suite 2, Hatfield, Pretoria
  - Sunninghill Clinic, Suite 3, Sunninghill

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the main FE200486 CS12 study were asked to continue into the FE200486 CS12A extension study.
Pre-assignment Details: 189 participants were randomized into the main study CS12 and 147 patients completed CS12. Of these, 137 participants were recruited into the extension study CS12A and 109 participants signed the informed consent for dose shift.
Groups:
- Degarelix 80 mg: Participants who completed the CS12 study in the Degarelix 80 mg arm continued that dose into the CS12A extension study. A protocol amendment in January 2006 changed the dosage to 160 mg (40 mg/mL) for all study participants.
- Degarelix 120 mg: Participants who completed the CS12 study in the Degarelix 120 mg arm continued that dose into the CS12A extension study. A protocol amendment in January 2006 changed the dosage to 160 mg (40 mg/mL) for all study participants.
- Degarelix 160 mg: Participants who completed the CS12 study in the Degarelix 160 mg arm continued that dose into the CS12A extension study. A protocol amendment in January 2006 changed the dosage to 160 mg (40 mg/mL) for all study participants.
Period: Overall Study
Arm/Group | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Started | 45 (Safety analysis set) | 48 | 44
Switched to 160 mg | 32 (A protocol amendment changed the dosage to 160 mg (40 mg/mL) for all participants) | 41 | 36
Completed | 16 (Participants ongoing at the time of study closure were considered to have completed the study) | 22 | 12
Not Completed | 29 | 26 | 32
Not completed — Adverse Event | 15 | 16 | 15
Not completed — Lack of Efficacy | 5 | 1 | 2
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 9 | 4 | 13
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Difficult to attend visits | 0 | 1 | 0
Not completed — No study drug available | 0 | 1 | 0
Not completed — Intermittent therapy required | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg | Total
Number analyzed (Participants) | 45 | 48 | 44 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.9) | 70.8 (6.3) | 72.4 (7.7) | 71.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 45 | 48 | 44 | 137
Race (NIH/OMB) [Count of Participants; unit: Participants] — Safety analysis set
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 3 | 0 | 3
    White | 45 | 44 | 44 | 133
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: kilogram] — Safety analysis set
  kilogram | 79.4 (15.9) | 79.1 (13.2) | 76.8 (12.4) | 78.4 (13.9)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] — Safety analysis set
  kilogram per square meter | 26.4 (4.5) | 26.4 (3.4) | 25.7 (3.4) | 26.2 (3.8)
Curative Intent [Number; unit: participants] — Safety analysis set. A curative intent of Yes refers to participants who have been castrated via radical prostatectomy or radiotherapy.
  participants
    Yes | 3 | 3 | 3 | 9
    No | 42 | 45 | 41 | 128
Gleason Score [Number; unit: participants] — Safety analysis set. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive. Gleason score for one patient in 160 mg group was missing.
  participants
    2-4 | 10 | 11 | 5 | 26
    5-6 | 18 | 22 | 16 | 56
    7-10 | 17 | 15 | 22 | 54
Stage of Prostate Cancer [Number; unit: participants] — Safety analysis set. Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localized | 10 | 14 | 8 | 32
    Locally advanced | 16 | 15 | 18 | 49
    Metastatic | 5 | 7 | 6 | 18
    Not classifiable | 14 | 12 | 12 | 38
Time since Prostate Cancer Diagnosis [Mean (Standard Deviation); unit: days] — Safety analysis set.
  days | 355 (645) | 227 (590) | 457 (1086) | 343 (798)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Markedly Abnormal Change in Vital Signs and Body Weight
Description: Vital signs and body weight included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight at the end of trial as compared to baseline. The table presents the number of participants in each group with normal baseline and markedly abnormal value post-baseline.
Time Frame: 5 years
Population: The data include data from participants participating in both the main study (FE200486 CS12) and the extension study FE200486 CS12A.
Measure: Number; unit: participants
Arm/Group | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 45 | 48 | 44
participants
  Diastolic blood pressure <=50 and decrease >=15 | 3 | 5 | 10
  Diastolic blood pressure >=105 and increase >=15 | 9 | 5 | 9
  Systolic blood pressure <=90 and decrease >=20 | 1 | 2 | 2
  Systolic blood pressure >=180 and increase >=20 | 4 | 9 | 8
  Heart rate <=50 and decrease >=15 | 3 | 5 | 5
  Heart rate >=120 and increase >=15 | 1 | 1 | 0
  Body weight decrease of >=7 percent | 4 | 10 | 8
  Body weight increase of >=7 percent | 18 | 19 | 14

2. Primary Outcome: Liver Function Tests
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) alanine aminotransferase (ALT) levels, aspartate aminotransferase levels, and bilirubin levels plus the number of participants who had ALT increases >3x ULN and ALT increases >3x ULN with concurrently increased bilirubin >1.5 ULN.
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 45 | 48 | 44
participants
  Abnormal alanine aminotransferase (ALAT) | 19 | 18 | 23
  Abnormal aspartate aminotransferase | 18 | 23 | 21
  Abnormal bilirubin | 8 | 11 | 3
  ALAT >3x upper limit of normal (ULN) | 3 | 3 | 3
  ALAT >3x ULN, bilirubin >1.5x ULN | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Description: Each patient's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the patient's Case Report Form.
Arm/Group | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Serious Adverse Events (participants affected / at risk) | 19/45 | 20/48 | 10/44
Other Adverse Events (participants affected / at risk) | 35/45 | 41/48 | 38/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 80 mg (N=45) | Degarelix 120 mg (N=48) | Degarelix 160 mg (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (10) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal defect (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Neurotrophic keratopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (8)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 4 (5) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Angiogram (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intravertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Acoustic neuroma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carcinoma in situ of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebovascular accident (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral circulatory failure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Monoplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraparesis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Post polio syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 1 (3) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (2)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 80 mg (N=45) | Degarelix 120 mg (N=48) | Degarelix 160 mg (N=44)
Anaemia (Blood and lymphatic system disorders) | 3 (6) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (5) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (3)
Cataract (Eye disorders) | 2 (4) | 2 (4) | 3 (4)
Constipation (Gastrointestinal disorders) | 7 (9) | 2 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (6) | 5 (5) | 6 (7)
Nausea (Gastrointestinal disorders) | 5 (7) | 1 (2) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Injection site pain (General disorders) | 6 (28) | 11 (22) | 13 (48)
Fatigue (General disorders) | 6 (8) | 3 (7) | 6 (9)
Pyrexia (General disorders) | 6 (7) | 3 (6) | 6 (11)
Injection site erythema (General disorders) | 3 (4) | 2 (4) | 9 (15)
Injection site nodule (General disorders) | 3 (7) | 5 (6) | 5 (5)
Injection site swelling (General disorders) | 0 (0) | 4 (9) | 6 (13)
Oedema peripheral (General disorders) | 4 (6) | 4 (6) | 2 (4)
Asthenia (General disorders) | 4 (4) | 2 (2) | 2 (2)
Injection site inflammation (General disorders) | 1 (1) | 3 (3) | 4 (4)
Chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 2 (2)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 3 (4)
Influenza (Infections and infestations) | 6 (8) | 9 (15) | 8 (9)
Urinary tract infection (Infections and infestations) | 4 (6) | 6 (11) | 4 (4)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2) | 5 (8)
Nasopharyngitis (Infections and infestations) | 2 (7) | 2 (4) | 4 (8)
Pneumonia (Infections and infestations) | 3 (3) | 2 (3) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (5) | 1 (1)
Prostatic specific antigen increased (Investigations) | 11 (12) | 8 (10) | 7 (9)
Weight increased (Investigations) | 7 (7) | 9 (10) | 7 (7)
Weight decreased (Investigations) | 3 (3) | 7 (9) | 8 (8)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 3 (3) | 5 (7)
Blood urea increased (Investigations) | 2 (4) | 2 (2) | 5 (5)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (6) | 3 (5)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 2 (3) | 3 (5)
Blood creatinine increased (Investigations) | 2 (3) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (4) | 2 (3)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 2 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (9) | 6 (8) | 9 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 7 (7) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (4) | 3 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (5)
Mylagia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 5 (8) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 2 (4)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4) | 4 (5)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3)
Haematuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 5 (7)
Nocturia (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Renal collic (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (4) | 1 (1) | 3 (3)
Prostatism (Reproductive system and breast disorders) | 3 (4) | 0 (0) | 2 (2)
Gynaecomastia (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3) | 8 (11)
Dyspnoea (Reproductive system and breast disorders) | 3 (3) | 3 (4) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 3 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 2 (3)
Hot flush (Vascular disorders) | 19 (27) | 18 (18) | 17 (20)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 3 (4)
Orthostatic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.